CLINICAL TRIAL: NCT04861324
Title: Effects of a Lifestyle Intervention on Gestational Diabetes Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nevada, Las Vegas (Other)
Responsible Party: Principal Investigator, Arpita Basu, Associate Professor, University of Nevada, Las Vegas
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1610677
Record Dates: First submitted 2021-04-22; First posted 2021-04-27 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2023-02

CONDITIONS: Gestational Diabetes; Type 2 Diabetes; Nutritional and Metabolic Disease
MeSH Terms: conditions — Diabetes, Gestational; Diabetes Mellitus, Type 2; Metabolic Diseases | interventions — Diet Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prenatal Care/Nutrition Education (No Intervention): Standard prenatal care with primary care physician with USDA-based federal guidelines
- Fruit/veggie + postprandial physical activity (Experimental): Nutrition education on increasing fruit and vegetable consumption and physical education on increasing postprandial physical activity for the duration from GDM diagnosis till delivery
  Interventions: Behavioral: Dietary Intervention

INTERVENTIONS:
Behavioral: Dietary Intervention — Increasing fruit and vegetable by two servings a day and at least 30 min a day of postprandial physical activity
  Arms: Fruit/veggie + postprandial physical activity

SUMMARY:
The purpose of this study is to investigate the effects of nutrition education focusing on colorful fruit and vegetable intake with after-meal physical activity guidance on glycemic control and complications in women with gestational diabetes and pre-gestational diabetes.

DETAILED DESCRIPTION:
Diabetes (high blood sugar) developed during pregnancy can be harmful to the mother as it can lead to delivery complications because of a large baby and increases risks of type 2 diabetes and heart disease in the mother and baby in later life. Thus, pregnancy is a critical time during the human lifespan to make effective dietary changes that are safe for both mother and the fetus and reduce risks of developing diabetes and pregnancy complications. Women at risk for gestational diabetes will be randomly assigned to the standard care or the nutrition education group. Blood draws and other biomedical measures will be collected at baseline and at end of the study before delivery.

ELIGIBILITY:
Inclusion Criteria:

* high risk for gestational diabetes
* willing to make lifestyle changes
* history of diabetes

Exclusion Criteria:

* carrying more than one fetus
* history of chronic conditions except diabetes and hypertension

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Females going through pregnancy and diagnosed with gestational diabetes
Enrollment: 45 (Actual)
Dates: Start 2021-04-28 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
Maternal glycemic control | 12 weeks
  Blood glycated hemoglobin
Maternal gestational weight gain | 12 weeks
  Body weight
Maternal medication usage | 12 weeks
  Glucose-lowering medications
Maternal Lipids | 12 weeks
  LDL-cholesterol and triglycerides

SECONDARY OUTCOMES:
Maternal inflammation | 12 weeks
  Adipokines, C-reactive protein
Maternal serum carotenoids | 12 weeks
  Carotenoids indicating fruit and vegetable consumption

CONTACTS AND LOCATIONS:
Overall Officials: Arpita Basu, PhD, Principal Investigator — University of Nevada at Las Vegas
Locations (1):
- UNLV School of Medicine MFM clinic, Las Vegas, Nevada, United States